CLINICAL TRIAL: NCT00857129
Title: Differentiated Birth Service- an Improvement?
Brief Title: Can Differentiated Birth Care Improve the Service?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Principal Investigator, Stine Bernitz, Midwife MSc PhD student, Ostfold Hospital Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3100
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Low Risk Birth; Births With Low Risk Factor
Keywords: "normal birth"; "birth outcome"; "low risk birth"; "low risk units"; If type of birth care unit have effect on birth outcome; Apgar score; breast feeding frequency; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): Low risk women with expected normal birth are being Randomized to The Midwife-led Unit, with low amount of intervention, No epidural is offered, no medical augmentation available, unless for the active phase of the second stage. If extended surveillance is necessary or if the birth no longer is considered to be normal and needs to be taken over by a doctor, the woman will be transferred to either the Normal Unit or the Special Unit
- 2 (Experimental): Low-risk women are randomised to this Low-risk maternal unit, The Normal Unit.The unit is organised for low-risk women with expected normal birth. The unit has access to extended surveillance, epidural and operative vaginal deliveries. If extended surveillance is necessary for a woman randomised to this unit, she does not have to be transferred to a higher level of care. Instrumental vaginal deliveries can be carried out at this unit.
  Interventions: Procedure: Normal Unit
- 3 (Experimental): Women with expected normal births are being randomised to this Special birth unit designed to take care of women before, under and after birth. The Special Unit cares for women with extended need for surveillance, but does also handle low-risk women.
  Interventions: Procedure: Special birth unit

INTERVENTIONS:
Procedure: Normal Unit — low-risk patients randomised to Normal Unit
  Other Names: Normal Unit, low-risk women
  Arms: 2
Procedure: Special birth unit — Low-risk women are randomised to the Special birth unit. Organised to take care of women with extended need for surveillance before, under and after birth.
  Other Names: Standard care unit: The Special Unit.
  Arms: 3

SUMMARY:
Prospective evaluation of birth complication in three differently staffed and equipped units in the same hospital.

DETAILED DESCRIPTION:
The study will include approximately 1000 normal births in a county hospital. The mothers are randomly assigned to one of three different maternal wards; one run by midwives, one normally equipped according to national standards for a county hospital and one prepared for complicated births. Endpoints are number of operative births and complications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mother, normal pregnancy, no prior operations on the uterus, no prior birth complications, no condition with negative effect on pregnancy or birth,one fetus in head position, spontaneously going into birth between week 36,1 and 41,6 of pregnancy,normal cardiotocograph test BMI of 32 or less, smoking no more than 10 cigarettes per day, wants to participate in the study and signs the consent form.

Exclusion Criteria:

* Any condition that has negative effect on the pregnancy or the birth, more than one fetus, all other positions than head position, induction of labor,pre term or post term birth, BMI of more than 32, smoking more than 10 cigarettes per day, does not want to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1111 (Actual)
Dates: Start 2006-09; Primary Completion 2010-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of operative deliveries | one week

SECONDARY OUTCOMES:
number of registered complications | one week

CONTACTS AND LOCATIONS:
Overall Officials: Pal Oian, PhD, Principal Investigator — University of Tromso, Norway
Locations (1):
- Ostfold Hospital Trust, Fredrikstad, Norway

REFERENCES:
- [Derived] Bernitz S, Oian P, Sandvik L, Blix E. Evaluation of satisfaction with care in a midwifery unit and an obstetric unit: a randomized controlled trial of low-risk women. BMC Pregnancy Childbirth. 2016 Jun 18;16(1):143. doi: 10.1186/s12884-016-0932-x. PMID 27316335